CLINICAL TRIAL: NCT05583552
Title: A Phase II Study Evaluating the Efficacy and Safety of Imetelstat in Patients With HR Myelodysplastic Syndromes or AML Failing HMA-based Therapy
Brief Title: Study to Evaluate Imetelstat in Patients With High-Risk MDS or AML Failing HMA-based Therapy
Acronym: IMpress
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GCP-Service International West GmbH (Industry)
Collaborators: Geron Corporation (Industry); Universitätsklinikum Leipzig (Other); Saint-Louis Hospital, Paris, France (Other); QIMR Berghofer Medical Research Institute (Other); Australasian Leukaemia and Lymphoma Group (Other); Groupe Francophone des Myelodysplasies (Other); German Myelodysplastic Syndrome Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMpress_001
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-06

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — imetelstat; GRN163L peptide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single-arm imetelstat (Experimental)
  Interventions: Drug: Imetelstat sodium

INTERVENTIONS:
Drug: Imetelstat sodium — Intravenous injection
  Other Names: GRN163L

SUMMARY:
The purpose of this study is to evaluate the efficacy, in terms of hematologic improvement, and safety of imetelstat in participants with high-risk (HR) myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) that is relapsed/refractory to hypomethylating agents (HMAs) treatment. Responding patients are eligible to continue treatment until loss of response/disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male and female ≥ 18 years at the first screening
* Must be able to adhere to the study visit schedule and other protocol requirements
* Initial diagnosis of AML or MDS according to WHO 2016 classification
* At least one cytopenia
* Failure to achieve complete or partial response or hematological improvement observed after at least six azacitidine monotherapy or four decitabine monotherapy based 4-week treatment cycles administered during the past two years OR Failure to achieve complete or partial response or hematological improvement observed after at least two 4-week treatment cycles with azacitidine plus venetoclax or with decitabine plus venetoclax during the past two years OR Relapse after initial complete or partial response or hematological improvement observed after at least six (azacitidine) or four (decitabine) based 4-week treatment cycles administered during the past two years OR Relapse after initial complete or partial response or hematological improvement observed after at least two 4-week treatment cycles with azacitidine plus venetoclax or with decitabine plus venetoclax during the past two years OR Intolerance to treatment with HMA-based therapy during the past two years
* Not eligible for allogeneic stem cell transplantation
* ≥ 5% bone marrow blasts at screening
* Off all other treatments for AML/MDS for at least 14 days; granulocyte colony-stimulating factor (G-CSF) and erythropoietin are allowed before and during the study as clinically indicated
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Biochemical laboratory test values must be within the defined limits.
* Availability of blood counts and transfusion events for previous 16 weeks
* Women of childbearing potential and practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies. For females, these restrictions apply for 3 months after the end of dosing.
* A woman of childbearing potential must have a negative serum or urine pregnancy test at screening and agree to be tested on day 1 of every cycle and at End of Treatment (EOT)
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control. For males, these restrictions apply for 3 months after the end of dosing
* Patients who are relapsed or refractory to, or not eligible for, therapy with approved and available FLT3 or IDH1/IDH2 inhibitors or other approved targeted therapies.

Exclusion Criteria:

* Chemotherapy within the 14 days prior to the first dose of imetelstat being administered (other than hydroxyurea)
* Participant has known allergies, hypersensitivity, or intolerance to imetelstat or its excipients (refer to the Investigators Brochure (IB))
* Participant has received an experimental or investigational drug or used an invasive investigational medical device within 30 days prior to day 1 of Cycle 1
* Prior treatment with imetelstat
* Prior history of intensive chemotherapy or hematopoietic stem cell transplant
* Major surgery within 4 weeks prior to day 1 of Cycle 1 (excluding the placement of vascular access and other minor surgical procedures)
* Diagnosed or treated for malignancy other than MDS or AML, except:

Malignancy treated with curative intent and with no known active disease present for 3 years before day 1 of Cycle 1 Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated cervical carcinoma in situ without evidence of disease

* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of day 1 of Cycle 1, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known history of human immunodeficiency virus (HIV) or any uncontrolled active systemic infection requiring IV antibiotics
* Active systemic hepatitis infection requiring treatment (carriers of hepatitis virus are permitted to enter the study), or known acute or chronic liver disease including cirrhosis
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the participant 's safety, interfere with the imetelstat metabolism, or put the study outcomes at undue risk; Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Females who are pregnant or are currently breastfeeding or planning to become pregnant while enrolled in this study or within 3 months after the end of dosing
* Participant is a man who plans to father a child while enrolled in this study or within 3 months after the end of dosing
* Other:

Participant is in custody by order of an authority or a court of law Participation in another interventional clinical study within the last 3 months prior to signing the Informed consent form (ICF) or simultaneous participation in other interventional clinical studies Previous assignment to treatment during this study Close affiliation with the investigator (e.g., a close relative) or persons working at the study site Participant is an employee of the sponsor or involved Contract Research Organization (CRO) Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the Participant's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall Hematological Response Rate of Participants after Treatment with Imetelstat | After 4 Months of Treatment
  The combined response assessment criteria for MDS and AML based on IWG 2018 criteria (MDS) and the criteria of the European LeukemiaNet (AML) will be used to define responders.
  The response rate is calculated as number of responders divided by the number of all participants of the analysis set.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, MD, Principal Investigator — Universitätsklinikum Leipzig
Locations (11):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Royal Brisbane and Women's Hospitals, Brisbane
  - Linear Clinical Research, Nedlands
- France (4):
  - CHU Nantes - Hôtel Dieu, Nantes
  - Hôpital Archet 1, Nice
  - Hôpital Saint-Louis, Paris
  - CHU de Toulouse, Toulouse
- Germany (4):
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universität Jena, Medizinische Fakultät, Jena
  - Universität Leipzig, Medizinische Fakultät, Leipzig
  - Klinikum rechts der Isar, München